CLINICAL TRIAL: NCT02517879
Title: Measuring Attendance of Community Point Distribution of Insecticide-treated Bed Nets and the Impact of Community Health Worker Hang-up in Rural Zambia: A Randomized Controlled Trial and Cost Analysis
Brief Title: Community Point Distribution of Insecticide Treated Bed Nets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDinsight (Other)
Collaborators: National Malaria Control Centre, Zambia (Unknown); Ministry of Health, Zambia (Other Government); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 003
Record Dates: First submitted 2015-07-27; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Malaria
Keywords: ITNs; malaria prevention
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 - 1-3 days (Experimental): Community health worker hang-up visit 1-3 days after the community point distribution
  Interventions: Other: Community point distribution; Other: Community health worker hang-up visit
- Group 2 - 5-7 days (Experimental): Community health worker hang-up visit 5-7 days after the community point distribution
  Interventions: Other: Community point distribution; Other: Community health worker hang-up visit
- Group 3 - 10-12 days (Experimental): Community health worker hang-up visit 10-12 days after the community point distribution
  Interventions: Other: Community point distribution; Other: Community health worker hang-up visit
- Group 4 - 15-17 days (Experimental): Community health worker hang-up visit 15-17 days after the community point distribution
  Interventions: Other: Community point distribution; Other: Community health worker hang-up visit
- Group 5 - No hang-up visit (Placebo Comparator): Did not receive any hang-up visit after the community point distribution
  Interventions: Other: Community point distribution

INTERVENTIONS:
Other: Community point distribution — Households were invited to a central location in their community (i.e. school, church, etc) where they received their allotment of ITNs (one per sleeping space, as pre-registered ahead of study activities). Households were provided with malaria prevention messaging at the distribution. They were called up one-by-one in front of other members of the community to mitigate misrepresentation of households.
Other: Community health worker hang-up visit — CHWs visited households to take stock of how many ITNs that were distributed during the distribution were hung and to hang any unhung ITNs.
  Arms: Group 1 - 1-3 days; Group 2 - 5-7 days; Group 3 - 10-12 days; Group 4 - 15-17 days

SUMMARY:
All households in three zones in Zambia's Eastern Province were invited to attend a community point distribution of insecticide treated bed nets (ITNs). Households were then randomized to different intervals for a community health worker (CHW) hang-up visit.

DETAILED DESCRIPTION:
Households were asked to attend a community point distribution of ITNs in one of three zones in Zambia's Eastern Province. Households that had been registered to receive ITNs were then randomized to one of five groups that received a CHW visit at different intervals. Group 1 was visited 1-3 days after distribution, group 2 was visited 5-7 days after, group 3 was visited 10-12 days after, group 4 was visited 15-17 days after, and group 5 did not receive a hang-up visit. Groups 1-4 were categorized as having received a hang-up visit and group 5 was categorized as not having received a hang-up visit. All households in all five groups were visited at 7-11 weeks after the distribution and again at 5-6 months after the distribution to assess short- and medium-term ITN retention and usage.

ELIGIBILITY:
Inclusion Criteria:

* Household was pre-registered by the National Malaria Control Centre to receive ITNs ahead of the start of study activities.
* Household was located in one of the three study areas of Mukonka, Lukwipa, and Chipeketi in Rufunsa District, Zambia

Exclusion Criteria:

* Household was not pre-registered to receive ITNs
* Household was not located in one of the three study areas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Community point distribution attendance | At time 0
  The percentage of pre-registered households that collected ITNs at the community point distributions on November 14, 19, and 21, 2013.
Self-installation of ITNs | Each group is randomized to receive a community health worker visit after a different duration, an average of 7 days after the point distribution
  The percentage of ITNs distributed to a household that the CHW found hanging at his/her visit.
Household ITN retention | An average of 9 weeks after community point distribution
  The percentage of ITNs distributed to a household that were found still in the household at the 7-11 week follow-up.
Household ITN retention | An average of 5.5 months after community point distribution
  The percentage of ITNs distributed to a household that were found still in the household at the 5-6 month follow-up.
Household percentage of ITNs hung | An average of 9 weeks after community point distribution
  The percentage of ITNs distributed to a household that were found hanging during the 7-11 week follow-up.
Household percentage of ITNs hung | An average of 5.5 months after community point distribution
  The percentage of ITNs distributed to a household that were found hanging during the 5-6 month follow-up.
Household percentage of sleeping spaces covered | An average of 9 weeks after community point distribution
  The percentage of sleeping spaces in the household that were covered by an ITN distributed during the community point distribution at the 7-11 week follow-up.
Household percentage of sleeping spaces covered | An average of 5.5 months after community point distribution
  The percentage of sleeping spaces in the household that were covered by an ITN distributed during the community point distribution at the 5-6 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, MPAID/MBA, Principal Investigator — IDinsight